CLINICAL TRIAL: NCT05249946
Title: FoodStep - a Sustainable Model for Food Services and Early Childhood Education and Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Suvi Virtanen (Other Government)
Collaborators: University of Helsinki (Other); Natural Resources Institute Finland (Other Government); Laurea University of Applied Sciences (Unknown)
Responsible Party: Sponsor-Investigator, Suvi Virtanen, Research Professor, Finnish Institute for Health and Welfare
Organization: Finnish Institute for Health and Welfare (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: THL/1646/6.00.00/2021
Record Dates: First submitted 2021-11-29; First posted 2022-02-22 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: Nutrition; Health; Food System; Sustainability; Children; Microbiome; Health Economics; Climate neutrality; Early childhood education; Food catering; Cost-effectiveness analysis
MeSH Terms: interventions — Food Services

STUDY DESIGN:
Intervention Model Description: Cluster-randomized Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): * increasing provision of vegetables and sustainable fish in food offered in early childhood education and care (ECEC) and adjusting intake of meat and milk to reasonable levels to meet recommendations
  * advancing food education, reducing food waste and assessing the climate and financial impacts of the shift towards a more plant-based diet
  Interventions: Other: FoodStep - a sustainable health-promoting model for food services and early childhood education and care
- Control group (No Intervention): Food supply and food education continue as usual.

INTERVENTIONS:
Other: FoodStep - a sustainable health-promoting model for food services and early childhood education and care — The investigators create a sustainable food system model that reduces the climate impact of the food system in early childhood education and care. In practice, the investigators i) promote plant-rich recipes, sustainable food purchases and consumption through municipality food services, ii) renew food education, and iii) reduce food waste in early education and care. To ensure the feasibility and long-term commitment, the investigators bring together municipal stakeholders and key actors within the food system and education sectors to co-create the content of a sustainable food system intervention. The randomized controlled intervention will be carried out at 26 daycare centers within four municipalities in Finland. The impact of the changes at a food system level on children's dietary intake and nutritional status, costs of the whole food system, the climate impact of the menus and children's diets as well as food waste in the daycare centers will be examined.
  Arms: Intervention group

SUMMARY:
Transformation towards a more climate-friendly and healthy sustainable diet will require major changes in the food system: increase in consumption of plant-based foods and only moderate consumption of animal-based foods. In the FoodStep -project, the investigators will develop a sustainable model for food system that reduces the climate impacts of the food system in early childhood education and care. The impact of the changes on children's nutrition, the climate impact of the diet, and the cost of food services will be assessed in a randomised controlled trial. In addition, the effects of the model on the knowledge and attitudes of decision-makers, experts in food service and early childhood education, and families are studied. Based on the project, the model can be applied nationally as part of Finland's climate change mitigation and adaptation strategy. Study aim to a sustainable food system reform through concrete guidelines, communication, and action initiatives.

ELIGIBILITY:
Inclusion Criteria:

* Are attending a full time daycare

Exclusion Criteria:

-

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change in daycare diet of the children | Before the intervention and 1 year after the intervention
  The investigators assess the change in vegetable, red meat and milk supply at daycare measured with Food Frequency Questionnaire.
Change in climate impact of Food System model at systemic level | Before the intervention and 1 year after the intervention
  The investigators assess the change in carbon footprint of daycare food supply.
Change in food service cost of Food System model at systemic level | Before the intervention and 1 year after the intervention
  The investigators assess how the costs change at food services due to the food system intervention and how cost-effective is the food system intervention compared to the food system as usual.
  Data comes from accounting of food services and book keeping: time spent to different tasks in food services.

CONTACTS AND LOCATIONS:
Locations (1):
- The Finnish Institute for Health and Welfare, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No